CLINICAL TRIAL: NCT02985086
Title: The Role of Antibiotic Prophylaxis in Immediate Versus Delayed Induction in Term-PROM - a Randomized Controlled Trial
Brief Title: Immediate Versus Delayed Induction in Term-PROM Using or Not Antibiotic Prophylaxis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Santa Maria, Portugal (Other)
Responsible Party: Principal Investigator, Filipa Faria Vaz Passos, Principal Investigator, Hospital de Santa Maria, Portugal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SantaMariaGarciadeOrtaPortugal
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Maternal Infection During Pregnancy (Diagnosis); Neonatal Infection
Keywords: term premature rupture of membranes, antibiotic prophylaxis, chorioamnionitis, endometritis, neonatal infection
MeSH Terms: conditions — Disease; Fetal Membranes, Premature Rupture; Chorioamnionitis; Endometritis | interventions — Cefoxitin; Oxytocin; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Immediate induction with antibiotic prophylaxis (Active Comparator): Immediate induction with antibiotic prophylaxis
  Interventions: Drug: Cefoxitin; Drug: oxytocin/misoprostol
- Immediate induction without antibiotic prophylaxis (Active Comparator): Immediate induction without antibiotic prophylaxis
  Interventions: Drug: oxytocin/misoprostol
- Delayed induction with antibiotic prophylaxis (Active Comparator): Delayed induction (>= 12 hours after PROM) with antibiotic prophylaxis
  Interventions: Drug: Cefoxitin; Drug: oxytocin/misoprostol

INTERVENTIONS:
Drug: Cefoxitin
  Arms: Delayed induction with antibiotic prophylaxis; Immediate induction with antibiotic prophylaxis
Drug: oxytocin/misoprostol

SUMMARY:
The primary aim of this study is to determine if antibiotics combined with immediate induction can significantly reduce the rate of maternal and neonatal infection compared with immediate induction alone in women presenting with PROM later than the 37+0 weeks of gestation. The secondary aim is to compare the rates of infection between immediate and delayed induction in women submitted to antibiotic prophylaxis.

DETAILED DESCRIPTION:
In a randomized controlled non-blind trial, low-risk women with singleton term pregnancies and a negative Group B Streptococcus culture presenting with PROM are randomly assigned to group A (immediate induction with antibiotic prophylaxis), group B (immediate induction without antibiotic prophylaxis) or group C (delayed induction with antibiotic prophylaxis).

ELIGIBILITY:
Inclusion Criteria:

* term (≥ 37+0 weeks) singleton pregnancy, a vertex presentation, ruptured membranes for less than 12 hours and a negative Group B Streptococcus (GBS) culture performed between 35 and 37 weeks.

Exclusion Criteria:

* active labor, absence of GBS culture or indication for GBS antibiotic prophylaxis, contraindication to expectant management or to vaginal delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 568 (Estimated)
Dates: Start 2013-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Maternal and neonatal infection rate | intrapartum and immediate postpartum

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Hospital Garcia de Orta, EPE, Almada
  - Hospital de Santa Maria, CHLN, EPE, Lisbon